CLINICAL TRIAL: NCT03279055
Title: Web-based Insomnia Treatment for Adolescent and Young Adult Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Alex's Lemonade Stand Foundation (Industry)
Responsible Party: Principal Investigator, Eric Zhou, Eric Zhou, PhD, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 17-276
Record Dates: First submitted 2017-09-09; First posted 2017-09-12 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Insomnia
Keywords: Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHUTi (Experimental): * Participants will be provided with an individual access code for SHUTi
  * SHUTi is delivered over 6 sessions, each taking 20-30 minutes
  * SHUTi is delivered by a virtual therapist
  * Participants will learn about the etiology and maintenance of their insomnia
  * Participants will learn how to maintain their sleep log
  * Participants will learn how to address lifestyle barriers that impact their sleep
  * Participants will be taught stimulus control techniques targeting non-sleep behaviors in the bedroom
  * Participants will learn a range of cognitive techniques that address the key cognitive factors that perpetuate poor sleep behavior
  * Participants will be taught how to gradually expand their restricted sleep
  Interventions: Behavioral: SHUTi

INTERVENTIONS:
Behavioral: SHUTi — Sleep Healthy Using the Internet (SHUTi) is a publicly available insomnia intervention program. It focuses on 5 treatment components that form the core of CBT-I: sleep restriction, stimulus control, cognitive restructuring, sleep behaviors, and relapse prevention.

SUMMARY:
This research study is evaluating a six-session online program designed to help insomnia (difficulty falling or staying asleep) in adolescent and young adult cancer survivors.

DETAILED DESCRIPTION:
The purpose of this study is to learn whether an adapted version of SHUTi (Sleep Healthy Using the Internet), a six-session online program which has been found to be effective in other groups of people, will be useful in treating insomnia in adolescent and young adult cancer survivors.

ELIGIBILITY:
Inclusion Criteria:

* 14-25 years of age
* History of a cancer diagnosis
* No active cancer therapy (excluding chemoprevention) in the past three months, and no cancer therapy currently planned in the next 6 months
* No surgery planned in the next 6 months
* Significant insomnia as evidenced by an Insomnia Severity Index score ≥12
* Able to read and write in English
* Has internet access at home
* Motivated and able to follow the demands of the SHUTi program, to keep sleep records, complete self-report symptom reports and make changes in their sleep schedule, including restricting their sleep

Exclusion Criteria:

* Prior attempt(s) to treat insomnia using cognitive-behavioral treatment for insomnia
* History of Bipolar Disorder diagnosis
* History of a Seizure Disorder diagnosis or have experienced a seizure in the past 12 months
* Intention to adjust (decrease or increase) use of sedative, hypnotic, or over-the-counter (e.g., Benadryl, Unisom) medications that can affect sleep during the study period
* Diagnosed, untreated sleep apnea or sleep apnea suspected by a physician but which has not been unevaluated, or other sleep disorder
* Employment that involves irregular sleep patterns, such as shift-work or frequent long-distance travel that involves adjusting to different time zones, or employment in a position that could impact public safety (such as operating heavy machinery)
* Refusal to modify or reduce excessive alcohol use that is likely to interfere with an individual's sleep

Ages: 14 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2018-08-10 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Insomnia symptoms | 8 weeks
  Insomnia symptom severity will be assessed using the Insomnia Severity Index

SECONDARY OUTCOMES:
Sleep efficiency | 6 weeks
  Sleep diary calculated sleep efficiency
Quality of life | 8 weeks
  Measured with PedsQL
Daytime sleepiness | 8 weeks
  Measured with Pediatric Daytime Sleepiness Scale

CONTACTS AND LOCATIONS:
Overall Officials: Eric Zhou, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhou ES, Recklitis CJ. Internet-delivered insomnia intervention improves sleep and quality of life for adolescent and young adult cancer survivors. Pediatr Blood Cancer. 2020 Sep;67(9):e28506. doi: 10.1002/pbc.28506. Epub 2020 Jun 22. PMID 32568460